CLINICAL TRIAL: NCT05805189
Title: Prospective Evaluation of Biophysical Parameters as Long-term Predictors of PVI With Multi-Electrode Radiofrequency Catheter: Comparison Between CARTO Guided and Fluoroscopy Guided Approach (MERCY Study)
Brief Title: Prospective Evaluation of Biophysical Parameters as Long-term Predictors of Pulmonary Vein Isolation
Acronym: MERCY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: MERCY
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, randomized study, designed to evaluate the acute achievement of pulmonary vein isolation with HELIOSTAR Balloon catheter. In this study, patients will be treat using prospectively the pre-ablation indicators of optimal electrode positioning in comparison with standard positioning evaluated by fluoroscopy visualization and contrast injection and the optimized biophysical parameters as predictors of long-term efficacy.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heliostar group A (Experimental): In this group the achievement of isolation of the pulmonary veins is evaluated with one shot tecnology Heliostar, multielecrode radiofrequency ballon catheter guided by the impedance level measured in the veins
  Interventions: Procedure: pulmonary vein (PV) isolation
- Carto Group B (Active Comparator): In this group the achievement of isolation of the pulmonary veins is evaluated with classic method guided by fluoroscopy
  Interventions: Procedure: pulmonary vein (PV) isolation

INTERVENTIONS:
Procedure: pulmonary vein (PV) isolation — The settings used during ablation will be for both groups: 15W, unipolar; 5ml/min baseline irrigation, 35ml/min irrigation during inflation/RF application; 55°C target electrode temperature; RF application time 60s for anterior electrodes, 20s for posterior electrodes. The catheter insertion in Pulmonary vein and ablation workflow will be different for two groups.

SUMMARY:
Current, worldwide assessments of the prevalence of AF estimate that 33 million people are affected by this cardiac arrhythmia. As the most common sustained atrial arrhythmia, AF has a well-established association with systemic embolic events, stroke, heart failure, and increased mortality. Current treatment guidelines and consensus statements for patients with AF suggest that most patients should be first managed with a pharmaceutical drug therapy; however, when a patient becomes drug refractory (intolerant or non-responsive), catheter ablation by PV isolation (PVI) is recommended.

The aim of PVI is abolishment of all conducted electrical activity beyond the isolating lesions.

The recent NICE guidelines have established that today RF point-by-point ablation is the most cost-effective treatment approach over a lifetime after failure of 1 or more anti-arrhythmic drugs5, but until now a new technology, HELIOSTAR, RF Balloon, has not been included in this cost-effectiveness analysis

DETAILED DESCRIPTION:
The multi-electrode RF Balloon catheter (HELIOSTAR, Biosense Webster) is a compliant Balloon with 10 circularly orientated electrodes bonded to its surface. It has been designed to be used in conjunction with the Carto3 system (Biosense Webster, CA). It is able to deliver RF energy directly forming a continuous circular ablation lesion around the PV ostia. With HELIOSTAR, each individual electrode can sense temperature and can be controlled separately. The electrodes can be used for visualization, stimulation, recording and ablation. The compliance of the Balloon allows conformation to the anatomy of the PVs and therefore maximizing tissue contact. The advantages of the RF Balloon include the ease of use to the operator that is associated with Balloon delivery systems, possibility of single shot PVI with tailored RF energy delivery, potentially shorter procedure times and avoidance of collateral damage to non-PVI structures, due to the capacity to individually select and deselect electrodes during ablation.6,7 To date, retrospective analyzes conducted in the RADIANCE and SHINE studies have shown the pre-ablation indicators of optimal electrode positioning and post-RF indicators associated with better outcomes; specifically, baseline impedance range 90-110 Ohms, impedance variability across ten electrodes ≤20 Ohms, baseline electrode temperature ≤31°C, baseline temperature variability ≤3°C and the post-RF indicators (impedance drop ≥12 Ohm and temperature rise ≥6°C) seem to independently predict a durable PVI. To the best of our knowledge, no studies have investigated prospectively the performance of impedance drop and temperature rise of HELIOSTAR ablation in terms of feasibility, acute PVI and post-procedural outcomes.

ELIGIBILITY:
Inclusion Criteria:

The following criteria must be met for subjects to be eligible for inclusion into the study

* Subjects indicated for the treatment of paroxysmal AF with the RF ablation system according to current and future Guidelines and system indications for use
* Subjects who are willing and capable of providing informed consent
* Patients who have stopped amiodarone for at least one month
* Subjects whose age is > 18 years old
* Subjects whose age is < 80 years old
* Subjects who are willing and capable of participating in all testing associated with this clinical study at an approved clinical investigational center

Exclusion Criteria:

Subjects who meet any one of the following criteria will be excluded from this clinical study

* Patients who had already undergo an AF ablation procedure
* Any known contraindication to an AF ablation or anticoagulation, including those listed in the instructions for use
* Subjects with indication for treatment of AF that is not according to current and future Guidelines and system indications for use
* Presence of an intracavitary thrombus
* Subjects that are unable or not willing to complete follow-up visits and examination for the duration of the study
* Patients with left ventricular ejection fraction < 35%
* Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon investigator's discretion)
* Hematological contraindications to ionizing radiation exposure
* Presence of complex congenital heart disease, and cardiac surgery within 1 month from enrollment
* Uncontrolled heart failure
* Subjects with severe valvular disease OR with a prosthetic - mechanical or biological- heart valve (not including valve repair and annular rings)
* Contraindications to general anesthesia
* Subjects who are currently enrolled in another investigational study or registry that would directly interfere with the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pulmonary vein single shot isolation | 12 months
  The primary objective of this study is PV single shot isolation in acute and at 1-3-6-12 months follow up with stringent monitoring including medical examination (Echo, ECG, and 24h-Holter)..
  It will be assessed the time necessary to reach the isolation, the number of erogations, the fluoroscopy dose and any use of contrast medium and they will be compared between the two arms.
  Our aim is to demonstrate that, even in the case of equivalent relapse rates during the follow up, the CARTO guided approach allows patients to benefit from a faster and less invasive procedure compared to the fluoroscopy guided method. This occurs because the former doesn't require contrast medium and the fluoroscopy time is notably reduced.

SECONDARY OUTCOMES:
Correlation of biophysical parameters, procedural, and ablation times | 12 months
  correlation of biophysical parameters, procedural, and ablation times between two groups. Therefore the following parameters will be collected: Balloonballoon dwelling time, impedance drop, and temperature rise of each RF sessions, rate of bonus and segmental applications, rate of reconnection. One of the endpoint is the recurrence of atrial tachycardia (AT) and AF after the blanking period (3 months), as measured by ECG and 24h-holter. It will be evaluated by the failure-free rate at 12 months post-index procedure in each cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Saverio Iacopino, MD, Principal Investigator — Maria Cecilia Hospital
Locations (1):
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: No
The Investigator must document in the subject's medical chart that informed consent has been obtained. The signed Informed Consent Form must be kept in the hospital/clinic medical chart or with the study subject documentation and be available for monitoring and auditing.